# Study of Asthma Phenotypes and Pharmacogenomic Interactions by Race-Ethnicity (SAPPHIRE)

Clinicaltrials.gov number: NCT01142947

Updated: September 19, 2016

(SAPPHIRE) - NCT01142947 Last updated: 02/19/2019

### **PROTOCOL**

# **Study population**

All SAPPHIRE individuals were recruited from Henry Ford Health System, whose Institutional Review Board approved this study. Informed written consent was obtained prior to the collection of any data. If the participant was a minor (age <18 years), informed written consent was obtained from a legal guardian and written assent was obtained from the participant. Individuals were eligible to participate as asthma cases if they were 12-56 years of age, had a documented physician diagnosis of asthma, and no prior diagnosis of congestive heart failure or chronic obstructive pulmonary disease.

At the time of enrollment, participants underwent a research evaluation. Lung function testing was performed using a pneumotachometer in accordance with 2005 ATS/ERS guideline recommendations. Reversible airway obstruction was assessed by administering 360µg (4 puffs) of albuterol sulfate from a standard metered dose inhaler (MDI). Spirometry was obtained before and 15 minutes after bronchodilator administration. For individuals with  $\leq$ 12% improvement in their forced expiratory volume at 1 second (FEV<sub>1</sub>), a second dose of albuterol (360µg for individuals  $\geq$ 18 years and 180µg for individuals <18 years) was administered followed by lung function reassessment 15 minutes after the second dose. Individuals were considered to have reversible airway obstruction if their FEV<sub>1</sub> improved by >12% after bronchodilator administration.

## **Discovery Group**

Study participants who met the following criteria were invited to undergo a 6-week course of inhaled beclomethasone dipropionate hydrofluoroalkane (beclomethasone HFA): no use of inhaled or systemic corticosteroids in the 4 weeks preceding the evaluation, a prebronchodilator FEV<sub>1</sub> that was 40-90% of predicted, reversible airway obstruction (i.e., >12% change in FEV<sub>1</sub> with albuterol administration), no smoking in the year prior to the evaluation and <10 pack-year smoking history in total, and not pregnant at the time of evaluation. Individuals who met these criteria and consented to undergo treatment were instructed to use 320µg (i.e., 2 puffs twice a day) of beclomethasone HFA daily via MDI (QVAR, Teva Respiratory LLC, Horsham, PA) with the use of a spacer device (AeroChamber Plus Flow-Vu spacer, Monaghan Medical Corp., Plattsburgh, NY). Treatment adherence was monitored using a DOSER-CT device (Meditrack, Easton, MA). This adherence monitoring device was fitted to each ICS MDI to count the total number of actuations. The group of individuals who completed the 6-week course of ICS treatment and had genome wide genotype data (described below) comprised the biomarker discovery group. Genome-wide genotyping was performed in African American individuals (self-reported race-ethnicity), who collectively comprised the largest population group in the SAPPHIRE cohort. As a result, the discovery sample consisted of 244 African American individuals who had both completed 6 weeks of study administered ICS treatment and genome-wide genotype data.

Genome-wide genotyping was performed using DNA isolated from whole blood and the Axiom AFR array (Affymetrix Inc., Santa Clara, CA). Quality control of the array results included a dish quality control measure  $\geq 0.82$ , an overall call rate  $\geq 97\%$ , and no discordance between patient-reported sex and the measured X-heterozygosity. Genotyped single nucleotide polymorphisms with an overall SNP call rate < 95%, a minor allele frequency (MAF) < 5%, or

(SAPPHIRE) - NCT01142947 Last updated: 02/19/2019

exact Hardy-Weinberg equilibrium p-value <10<sup>-4</sup> were removed from the analysis. Only autosomal SNPs were analyzed.

# Validation Groups

Validation was carried out in 2 additional groups from the SAPPHIRE cohort. The primary validation set consisted of African American SAPPHIRE participants (n=803) who met the following criteria: available prospective clinical data on asthma exacerbations from available electronic health records, measures of ICS exposure through pharmacy claims records, existing genome-wide genotype data meeting QC standards, and African American race-ethnicity by participant self-report. Health records were used to identify severe asthma exacerbations and generate measures of ICS exposure over time. Severe asthma exacerbation were defined as those requiring burst oral corticosteroids, an emergency department visit, or a hospitalization.

We standardized each available ICS preparation on the U.S. market by multiplying the number of actuations per container by the milligram dose released per actuation and dividing by the milligram strength of the lowest recommended dose for that preparation as specified in National Asthma Education and Prevention Program. Expert Panel Report 3 (ERP-3) guidelines. Applying our standardization method to participant health data, we assigned each prescription fill the value assigned for each preparation and divided by the total number of days between fills (i.e., days until the next fill) to approximate the amount of ICS used each day. We summed each daily value for 6 months and and divided by 180 to create a measure that could be interpreted as a 6-month average of the daily number of ICS doses (in units of what ERP-3 guidelines defined as a "low" dose for that preparation). This process was repeated for each day of each individual's follow-up to create a moving window of ICS exposure for participant in the primary validation set. We also created a dichotomous indicator variable for each day of follow-up to denote when a patient had used a long-acting beta-agonist (LABA) in the preceding 180 days. As time-updated proxy measures of asthma severity, we created separate exposure variables for short-acting beta-agonist (SABA) MDI and nebulizer use. The SABA measures were calculated by summing the doses filled over a 90 day moving window. Therefore, the SABA measures represented the average number of SABA doses used per day in the preceding 3-months. We also created a baseline asthma severity measure based on asthma rescue medication use in the preceding year as described by Allen-Ramey et al. (J Manag Care Pharm 2006; 12:310-21).

The second validation group comprised European American individuals from the SAPPHIRE cohort (n=98) who met the same selection criteria and underwent the same 6-week ICS treatment protocol as the discovery set. Because this group of European American SAPPHIRE participants had the same treatment regimen and follow-up duration as the discovery set, change in ACT composite score was used as the outcome variable. Participants in this second validation group were genotyped for the rs3827907 SNP using a TaqMan SNP Genotyping Assay (Applied Biosystems).

### **Statistical Analysis**

In the discovery analysis, we used an additive genetic model and linear regression to assess the relationship between genotype and change in ACT score over 6 weeks of ICS treatment. To capture both an independent genetic effect and a modifying effect on ICS treatment response, we included both the main effect of each SNP and an interaction term between the SNP and ICS exposure. The full model also included individual variables for patient age, sex, ACT score at

(SAPPHIRE) - NCT01142947 Last updated: 02/19/2019

baseline (i.e., the time of enrollment into the study), smoking status (coded as never, past, and present), the first three principal components (derived using the program EIGENSOFT and representing underlying population substructure), and ICS exposure (continuous measure based on adherence). To jointly test the effect of the SNP and the SNP x ICS interaction, we compared the full model containing all of the aforementioned variables with a reduced model (i.e., all of the variables in the full model except for the SNP and interaction term) using an F-test.

SNP associations with P<5.0x10<sup>-7</sup> (strict Bonferroni correction P<0.05/574,370=8.71x10<sup>-8</sup>) from the discovery were reassessed in the validation groups. The primary validation analysis was performed in African American SAPPHIRE participants who were not involved in the 6 weeks of study-administered ICS treatment but did have longitudinal clinical information on asthma exacerbations (n=803). Proportional hazards regression was used to evaluate the association between both the SNP term and the SNP x ICS interaction term with time-to-severe asthma exacerbation. These models also accounted for patient age, sex, BMI, smoking status, ACT score at baseline (i.e., enrollment), baseline asthma severity score, LABA use (an indicator variable denoting use of an ICS-LABA combination inhaler), time-updated measures of SABA MDI and nebulizer use, the first 3 principal components, and the time-updated ICS exposure measure. A 2-degree of freedom likelihood ratio test was used to evaluate the significance of the difference in model fit for all variables as compared with a reduced model without the SNP and the SNP x ICS interaction terms.

We also assessed for replication in the 98 European American SAPPHIRE participants who completed 6-weeks of ICS treatment. The linear regression analysis was the same as used in the discovery set with the exception that only the top variant, rs3827907, was assessed, and the regression model did not include principal components to account for underlying population structure.

Analyses were performed using R statistical software.

(SAPPHIRE) - NCT01142947 Last updated: 02/19/2019

#### FIGURE LEGENDS

Figure E1. Quantile-quantile (Q-Q) plot of expected vs. observed genome-wide joint association test results before (A) and after (B) applying genomic control. Each joint test estimated the combined effect of a single nucleotide polymorphism (SNP) and its interaction with inhaled corticosteroid (ICS) use on changes in asthma control occurring over 6 weeks of ICS treatment. Asthma control was measured using the composite Asthma Control Test (ACT) score. The models also adjusted for patient age, sex, ACT score at baseline (i.e., the time of study enrollment), smoking status, the first three principal components, and ICS adherence. The Q-Q plot before applying genomic control (plot A) showed mild inflation ( $\lambda$ =1.09); this was corrected via genomic control (plot B).

Figure E2. LocusZoom plot of rs3827907 on chromosome 14. Single nucleotide polymorphisms located within a 200 kilobase window upstream and downstream of rs3827907 are shown. P-values were generated using the joint (SNP and SNP\*ICS combined) test of association with changes in asthma control occurring over 6 weeks of ICS treatment. The SNP color represents the level of correlation between each SNP and rs3827907. Genes located in the region are shown beneath the plotted SNPs.

Figure E3. Relationship between rs3827907 genotype and absolute change in Asthma Control Test (ACT) composite score among African American participants in the Study of Asthma Phenotypes and Pharmacogenomic Interactions by Race-ethnicity (SAPPHIRE) following 6 weeks of observed inhaled corticosteroid (ICS) treatment. Results are restricted to the 129 individuals whose asthma was not controlled at baseline (ACT score ≤19) and are stratified by levels of patient ICS use (≤75% adherence was considered low use and >75% adherence was considered high use). Black lines connect the means for each group.

Figure E4. Relationship between rs3827907 genotype and absolute change in Asthma Control Test (ACT) composite score among African American participants in the SAPPHIRE cohort following 6 weeks of observed inhaled corticosteroid (ICS) treatment (n=244). The rs3827907 genotype is categorized in TT homozygotes and C-allele carriers (denoted C- and representing individuals with either the CT or CC genotypes). Results are stratified by levels of patient ICS use (≤75% adherence was considered low use and >75% adherence was considered high use). Black lines connect the means for each group.

Figure E5. Relationship between rs3827907 genotype and absolute change in Asthma Control Test (ACT) composite score among European American participants in the Study of Asthma Phenotypes and Pharmacogenomic Interactions by Race-ethnicity (SAPPHIRE) cohort following 6 weeks of observed inhaled corticosteroid (ICS) treatment (n=98). Results are stratified by levels of patient ICS use (≤75% adherence was considered low use and >75% adherence was considered high use). Black lines connect the means for each group.

Figure E6. Correlation of expression between protein-coding genes located within 1 megabase upstream and downstream of rs3827907 on chromosome 14. Gene expression is based on read counts from RNA-seq data obtained from 158 African American participants from the Study of

(SAPPHIRE) - NCT01142947 Last updated: 02/19/2019

Asthma Phenotypes and Pharmacogenomic Interactions by Race-ethnicity (SAPPHIRE). Read counts were normalized using the program DESeq2

(https://bioconductor.org/packages/release/bioc/html/DESeq2.html). Gene expression of *EDDM3B* in whole blood was low and did not meet our criterion for evaluation (≥50% of individuals with read counts >0); therefore, it is not listed among the 32 genes evaluated for this region.

Figure E7. Effect of baseline measures of eosinophil-derived neurotoxin (EDN) on the relationship between rs3827907 C-allele carrier status and absolute change in Asthma Control Test (ACT) composite score among European American participants in the SAPPHIRE cohort following 6 weeks of observed inhaled corticosteroid (ICS) treatment (n=96). Results are stratified by levels of patient ICS use (≤75% adherence was considered low use and >75% adherence was considered high use) and pre-treatment serum levels of EDN. Low and high EDN levels were defined as those ≤2.34 ng/mL and >2.34 ng/mL, respectively. Black lines connect the means for each group.

Figure E8. Effect of baseline blood eosinophil counts on relationship between rs3827907 C-allele carrier status and absolute change in Asthma Control Test (ACT) composite score among European American participants in the SAPPHIRE cohort following 6 weeks of observed inhaled corticosteroid (ICS) treatment (n=94). Results are stratified by levels of patient ICS use ( $\leq$ 75% adherence was considered low use and  $\geq$ 75% adherence was considered high use) and blood eosinophil counts measured before ICS treatment. Low and high eosinophil counts were defined as those  $\leq$ 222 cells/ $\mu$ L and  $\geq$ 222 cells/ $\mu$ L, respectively. Black lines connect the means for each group.

Figure E9. LocusZoom plot of rs3827907 on chromosome 14 including imputed variants. Single nucleotide polymorphisms located within a 200 kilobase window upstream and downstream of rs3827907 are shown. P-values were generated using the joint (SNP and SNP\*ICS combined) test of association with changes in asthma control occurring over 6 weeks of ICS treatment. The SNP color represents the level of correlation between each SNP and rs3827907. After res3827907, the next most significant variant, imputed SNP rs12891518, is also labeled. Genes located in the region are shown beneath the plotted SNPs.

(SAPPHIRE) - NCT01142947 Last updated: 02/19/2019

### SUPPLEMENTAL REFERENCES

- 1. Miller MR, Crapo R, Hankinson J, Brusasco V, Burgos F, Casaburi R, et al. General considerations for lung function testing. Eur Respir J 2005; 26:153-61.
- 2. Miller MR, Hankinson J, Brusasco V, Burgos F, Casaburi R, Coates A, et al. Standardisation of spirometry. Eur Respir J 2005; 26:319-38.
- 3. Hankinson JL, Odencrantz JR, Fedan KB. Spirometric reference values from a sample of the general U.S. population. Am J Respir Crit Care Med 1999; 159:179-87.
- 4. Bender B, Wamboldt FS, O'Connor SL, Rand C, Szefler S, Milgrom H, et al. Measurement of children's asthma medication adherence by self report, mother report, canister weight, and Doser CT. Ann Allergy Asthma Immunol 2000; 85:416-21.
- 5. O'Connor SL, Bender BG, Gavin-Devitt LA, Wamboldt MZ, Milgrom H, Szefler S, et al. Measuring adherence with the Doser CT in children with asthma. J Asthma 2004; 41:663-70.
- 6. Ewels P, Magnusson M, Lundin S, Kaller M. MultiQC: summarize analysis results for multiple tools and samples in a single report. Bioinformatics 2016; 32:3047-8.
- 7. Dobin A, Davis CA, Schlesinger F, Drenkow J, Zaleski C, Jha S, et al. STAR: ultrafast universal RNA-seq aligner. Bioinformatics 2013; 29:15-21.
- 8. Wang L, Wang S, Li W. RSeQC: quality control of RNA-seq experiments. Bioinformatics 2012; 28:2184-5.
- 9. Ramirez F, Dundar F, Diehl S, Gruning BA, Manke T. deepTools: a flexible platform for exploring deep-sequencing data. Nucleic Acids Res 2014; 42:W187-91.
- 10. Li B, Dewey CN. RSEM: accurate transcript quantification from RNA-Seq data with or without a reference genome. BMC Bioinformatics 2011; 12:323.
- 11. Love MI, Huber W, Anders S. Moderated estimation of fold change and dispersion for RNA-seq data with DESeq2. Genome Biol 2014; 15:550.
- 12. Reddel HK, Taylor DR, Bateman ED, Boulet LP, Boushey HA, Busse WW, et al. An official American Thoracic Society/European Respiratory Society statement: asthma control and exacerbations: standardizing endpoints for clinical asthma trials and clinical practice. Am J Respir Crit Care Med 2009; 180:59-99.
- 13. Williams LK, Peterson EL, Wells K, Ahmedani BK, Kumar R, Burchard EG, et al. Quantifying the proportion of severe asthma exacerbations attributable to inhaled corticosteroid nonadherence. J Allergy Clin Immunol 2011; 128:1185-91.
- 14. Wells KE, Peterson EL, Ahmedani BK, Severson RK, Gleason-Comstock J, Williams LK. The relationship between combination inhaled corticosteroid and long-acting beta-agonist use and severe asthma exacerbations in a diverse population. J Allergy Clin Immunol 2012; 129:1274-9.
- 15. Williams LK, Joseph CL, Peterson EL, Wells K, Wang M, Chowdhry VK, et al. Patients with asthma who do not fill their inhaled corticosteroids: a study of primary nonadherence. J Allergy Clin Immunol 2007; 120:1153-9.
- 16. Expert Panel Report 3 (EPR-3): Guidelines for the Diagnosis and Management of Asthma-Summary Report 2007. J Allergy Clin Immunol 2007; 120:S94-138.
- 17. Paris J, Peterson EL, Wells K, Pladevall M, Burchard EG, Choudhry S, et al. Relationship between recent short-acting beta-agonist use and subsequent asthma exacerbations. Ann Allergy Asthma Immunol 2008; 101:482-7.

(SAPPHIRE) - NCT01142947 Last updated: 02/19/2019

18. Allen-Ramey FC, Bukstein D, Luskin A, Sajjan SG, Markson LE. Administrative claims analysis of asthma-related health care utilization for patients who received inhaled corticosteroids with either montelukast or salmeterol as combination therapy. J Manag Care Pharm 2006; 12:310-21.

- 19. Nishimura KK, Galanter JM, Roth LA, Oh SS, Thakur N, Nguyen EA, et al. Early-life air pollution and asthma risk in minority children. The GALA II and SAGE II studies. Am J Respir Crit Care Med 2013; 188:309-18.
- 20. Neophytou AM, White MJ, Oh SS, Thakur N, Galanter JM, Nishimura KK, et al. Air Pollution and Lung Function in Minority Youth with Asthma in the GALA II (Genes-Environments and Admixture in Latino Americans) and SAGE II (Study of African Americans, Asthma, Genes, and Environments) Studies. Am J Respir Crit Care Med 2016; 193:1271-80.
- 21. Pino-Yanes M, Gignoux CR, Galanter JM, Levin AM, Campbell CD, Eng C, et al. Genome-wide association study and admixture mapping reveal new loci associated with total IgE levels in Latinos. J Allergy Clin Immunol 2015; 135:1502-10.
- 22. White MJ, Risse-Adams O, Goddard P, Contreras MG, Adams J, Hu D, et al. Novel genetic risk factors for asthma in African American children: Precision Medicine and the SAGE II Study. Immunogenetics 2016; 68:391-400.
- 23. Yang JJ, Li J, Buu A, Williams LK. Efficient inference of local ancestry. Bioinformatics 2013; 29:2750-6.
- 24. Choudhry S, Coyle NE, Tang H, Salari K, Lind D, Clark SL, et al. Population stratification confounds genetic association studies among Latinos. Hum Genet 2006; 118:652-64.
- 25. Yaeger R, Avila-Bront A, Abdul K, Nolan PC, Grann VR, Birchette MG, et al. Comparing genetic ancestry and self-described race in african americans born in the United States and in Africa. Cancer Epidemiol Biomarkers Prev 2008; 17:1329-38.
- 26. Price AL, Patterson NJ, Plenge RM, Weinblatt ME, Shadick NA, Reich D. Principal components analysis corrects for stratification in genome-wide association studies. Nat Genet 2006; 38:904-9.
- 27. Price AL, Zaitlen NA, Reich D, Patterson N. New approaches to population stratification in genome-wide association studies. Nat Rev Genet 2010; 11:459-63.
- 28. consortium Tgp. A map of human genome variation from population-scale sequencing. Nature 2010; 467:1061-73.
- 29. Alexander DH, Novembre J, Lange K. Fast model-based estimation of ancestry in unrelated individuals. Genome Res 2009; 19:1655-64.
- 30. Pino-Yanes M, Thakur N, Gignoux CR, Galanter JM, Roth LA, Eng C, et al. Genetic ancestry influences asthma susceptibility and lung function among Latinos. J Allergy Clin Immunol 2015; 135:228-35.
- 31. Consortium TIH. A second generation human haplotype map of over 3.1 million SNPs. Nature 2007:851-61.
- 32. Kraft P, Yen YC, Stram DO, Morrison J, Gauderman WJ. Exploiting gene-environment interaction to detect genetic associations. Hum Hered 2007; 63:111-9.
- 33. Fagny M, Paulson JN, Kuijjer ML, Sonawane AR, Chen CY, Lopes-Ramos CM, et al. Exploring regulation in tissues with eQTL networks. Proc Natl Acad Sci U S A 2017; 114:E7841-E50.

(SAPPHIRE) - NCT01142947 Last updated: 02/19/2019

34. Yao C, Joehanes R, Johnson AD, Huan T, Liu C, Freedman JE, et al. Dynamic Role of trans Regulation of Gene Expression in Relation to Complex Traits. Am J Hum Genet 2017; 100:571-80.

- 35. Stegle O, Parts L, Piipari M, Winn J, Durbin R. Using probabilistic estimation of expression residuals (PEER) to obtain increased power and interpretability of gene expression analyses. Nat Protoc 2012; 7:500-7.
- 36. R Core Team. R: A language and environment for statistical computing. Vienna, Austria: R Foundation for Statistical Computing, 2014.

Table E1. Interactions between previously reported pharmacogenetic variants and inhaled corticosteroid use on changes in

asthma control among individuals in the discovery set (n=244)\*

| SNP | Chr | Position | Imputation<br>Quality† | Allele‡ | MAF‡ | Gene | Parameter<br>estimate for<br>SNP§ | P-value for<br>SNP term | Parameter estimate for SNP x ICS interaction§ | P-value for interaction term | P-value for joint test¶ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| rs10044254 | 5 | 15,783,596 | 0.96 | G/A | 0.35 | FBXL7 | 2.49 | 0.060 | -3.08 | 0.063 | 0.167 |
| rs2395672 | 6 | 37,428,577 | 0.75 | A/G | 0.03 | CMTR1 | 2.38 | 0.583 | -1.72 | 0.750 | 0.566 |
| rs6924808 | 6 | 98,358,575 | 0.95 | G/A | 0.39 | | 0.41 | 0.733 | -0.70 | 0.651 | 0.861 |
| rs6456042 | 6 | 166,534,742 | 0.96 | A/C | 0.35 | T | 1.18 | 0.369 | -1.33 | 0.413 | 0.657 |
| rs3127412 | 6 | 166,535,561 | 0.96 | C/T | 0.35 | T | 1.18 | 0.369 | -1.33 | 0.413 | 0.657 |
| rs37972 | 7 | 8,007,509 | 0.92 | T/C | 0.18 | GLCCI1 | -0.20 | 0.910 | 0.44 | 0.840 | 0.918 |
| rs2691529 | 7 | 77,803,275 | 0.89 | C/T | 0.24 | MAGI2 | -0.86 | 0.564 | 0.77 | 0.685 | 0.713 |
| rs6467778 | 7 | 138,178,222 | 0.95 | A/G | 0.17 | TRIM24 | -1.43 | 0.354 | 1.36 | 0.481 | 0.521 |
| rs10481450 | 8 | 9,798,246 | 0.80 | A/T | 0.13 | | 2.88 | 0.092 | -2.63 | 0.248 | 0.061 |
| rs3793371 | 8 | 144,664,299 | 0.97 | A/G | 0.04 | EEF1D<br>(NAPRT1) | 2.03 | 0.761 | -2.32 | 0.760 | 0.954 |
| rs4271056 | 9 | 38,232,043 | 1.00 | C/T | 0.23 | , | -2.10 | 0.106 | 2.86 | 0.087 | 0.230 |
| rs7850103 | 9 | 118,137,835 | 0.99 | A/C | 0.15 | DEC1 (TNC) | 2.14 | 0.263 | -3.57 | 0.132 | 0.126 |
| rs1353649 | 11 | 20,253,599 | 0.99 | A/G | 0.40 | , | -1.45 | 0.203 | 2.31 | 0.113 | 0.194 |
| rs4980524 | 11 | 63,959,259 | 0.99 | C/A | 0.29 | STIP1 | 0.38 | 0.736 | -0.82 | 0.563 | 0.655 |
| rs6591838 | 11 | 63,959,356 | 0.99 | G/A | 0.21 | STIP1 | 0.43 | 0.736 | -0.53 | 0.744 | 0.944 |
| rs2236647 | 11 | 63,964,605 | 0.99 | C/T | 0.28 | STIP1 | -1.03 | 0.452 | 1.15 | 0.494 | 0.740 |
| rs1144764 | 11 | 77,870,486 | 0.94 | T/C | 0.39 | KCTD21-AS1<br>(ALG8) | -1.75 | 0.191 | 2.38 | 0.161 | 0.367 |
| rs12891009 | 14 | 74,083,846 | 0.93 | T/C | 0.26 | ACOT6/HEAT<br>R4 (ACOT4) | -0.18 | 0.884 | -0.24 | 0.877 | 0.580 |
| rs2230155 | 15 | 59,510,189 | 0.90 | A/G | 0.41 | MYO1E | 0.84 | 0.448 | -1.38 | 0.341 | 0.550 |
| rs12438740 | 15 | 59,515,767 | 1.00 | A/G | 0.41 | MYO1E | 0.58 | 0.601 | -0.97 | 0.507 | 0.744 |
| rs242941 | 17 | 43,892,520 | 1.00 | C/A | 0.37 | CRHR1 | 0.16 | 0.883 | 0.00 | 0.999 | 0.880 |
| rs242939 | 17 | 43,895,579 | 1.00 | C/T | 0.32 | CRHR1 | 2.19 | 0.081 | -2.82 | 0.085 | 0.215 |
| rs1876828 | 17 | 43,911,525 | 0.99 | T/C | 0.03 | CRHR1 | 5.29 | 0.459 | -5.67 | 0.497 | 0.701 |
| rs2240017 | 17 | 45,810,919 | 0.38 | G/C | 0.01 | TBX21 | 4.87 | 0.916 | -3.57 | 0.963 | 0.560 |
| rs1380657 | 17 | 48,598,785 | 1.00 | G/A | 0.12 | MYCBPAP<br>(SPATA20) | 2.95 | 0.113 | -4.70 | 0.052 | 0.081 |
| rs6504666 | 17 | 48,601,328 | 1.00 | G/A | 0.16 | MYCBPAP<br>(SPATA20) | 0.99 | 0.544 | -1.21 | 0.565 | 0.831 |
| rs9303988 | 18 | 6,667,583 | 0.67 | T/C | 0.44 | | 1.10 | 0.348 | -1.29 | 0.397 | 0.631 |
| rs279728 | 20 | 45,080,421 | 1.00 | T/C | 0.23 | | 0.75 | 0.551 | -0.98 | 0.538 | 0.826 |
| rs2037925 | 21 | 40,699,931 | 0.95 | C/T | 0.33 | (BRWD1) | -2.27 | 0.098 | 2.38 | 0.155 | 0.192 |
| rs2836987 | 21 | 40,706,594 | 0.94 | C/T | 0.31 | (BRWD1) | -1.53 | 0.272 | 1.65 | 0.334 | 0.503 |
| rs138335 | 22 | 41,227,086 | 0.83 | C/G | 0.07 | ST13 | 1.30 | 0.652 | -2.64 | 0.456 | 0.350 |
| rs138337 | 22 | 41,231,053 | 0.94 | G/A | 0.42 | ST13 | 0.79 | 0.504 | -1.09 | 0.465 | 0.759 |

SNP denotes single nucleotide polymorphism; Chr, chromosome; MAF, minor allele frequency; and ICS, inhaled corticosteroid. \*SNPs were selected from variants previously reported to be associated with ICS response. The outcome phenotype was the change in asthma control test (ACT) score from before to immediately following 6 weeks of inhaled corticosteroid (ICS) treatment. †The imputation quality score is the MACH-based imputation r² value, which ranges from zero to one. Values closer to one indicate higher imputation quality.

‡The "effect" allele is shown first, and the referent allele follows. The allele frequency of the "effect" allele is provided, and in the current table, this estimate is based on the observed frequency in the discovery set.

§The parameter estimates demonstrate the direction and magnitude for a change in the ACT score over the course of 6 weeks of ICS treatment. A *positive* parameter estimate indicates that the variable was associated with an improvement in asthma control over the course of treatment. The parameter estimate for the SNP can be interpreted as the effect on asthma control for each additional "effect" allele (i.e., none [=0], one [=1], or two alleles [=2]). The parameter estimate for the interaction term can be interpreted as the combined effect of increasing ICS use (i.e., going from zero to complete adherence to the prescribed dose [a continuous variable ranging from 0 to 1]) and the number of "effect" alleles on the change in asthma control over 6 weeks of ICS treatment.

The P-values for the SNP and SNP x ICS interaction variables are shown for the model simultaneously including these variables, as well as adjusting for patient age, sex, ACT score at baseline enrollment into the study, smoking status (coded as never, past, and present), the first three principal components, and ICS adherence.

¶The F-test assessed the significance of the difference in model fit between the full model (i.e., all of the aforementioned variables included) and the reduced model (i.e., the full model minus both the SNP and SNP x ICS interaction terms). In other words, a *joint test* was used to simultaneously assess the combined significance of the SNP and SNP x ICS interaction terms.

Table E2. Interactions between previously reported pharmacogenetic variants and inhaled corticosteroid use on severe

asthma exacerbations among African American SAPPHIRE participants in the validation set (n=803)\*

| SNP | Chr | Position | Imputation<br>Quality† | Allele‡ | MAF‡ | Gene | Parameter estimate for SNP§ | P-value<br>for SNP<br>term | Parameter estimate for SNP x ICS interaction§ | P-value for interaction term | P-value<br>for joint<br>test¶ |
|---|---|---|---|---|---|---|---|---|---|---|---|
| rs10044254 | 5 | 15,783,596 | 0.96 | G/A | 0.34 | FBXL7 | -0.18 | 0.115 | 0.13 | 0.433 | 0.282 |
| rs2395672 | 6 | 37,428,577 | 0.75 | A/G | 0.04 | CMTR1 | 0.28 | 0.326 | -0.88 | 0.036 | 0.020 |
| rs6924808 | 6 | 98,358,575 | 0.95 | G/A | 0.42 | | 0.00 | 0.981 | -0.18 | 0.212 | 0.331 |
| rs6456042 | 6 | 166,534,742 | 0.96 | A/C | 0.36 | T | 0.10 | 0.367 | 0.09 | 0.524 | 0.294 |
| rs3127412 | 6 | 166,535,561 | 0.96 | C/T | 0.36 | T | 0.10 | 0.367 | 0.09 | 0.524 | 0.294 |
| rs37972 | 7 | 8,007,509 | 0.92 | T/C | 0.21 | GLCCI1 | 0.20 | 0.104 | -0.22 | 0.188 | 0.233 |
| rs2691529 | 7 | 77,803,275 | 0.89 | C/T | 0.26 | MAGI2 | 0.16 | 0.154 | -0.04 | 0.742 | 0.336 |
| rs6467778 | 7 | 138,178,222 | 0.95 | A/G | 0.16 | TRIM24 | -0.40 | 0.017 | 0.21 | 0.304 | 0.039 |
| rs10481450 | 8 | 9,798,246 | 0.80 | A/T | 0.13 | | 0.13 | 0.437 | 0.07 | 0.717 | 0.508 |
| rs3793371 | 8 | 144,664,299 | 0.97 | A/G | 0.04 | EEF1D<br>(NAPRT1) | -0.71 | 0.016 | -0.29 | 0.361 | 3.27x10 |
| rs4271056 | 9 | 38,232,043 | 1.00 | C/T | 0.22 | , | 0.07 | 0.587 | 0.16 | 0.319 | 0.316 |
| rs7850103 | 9 | 118,137,835 | 0.99 | A/C | 0.11 | DEC1 (TNC) | 0.77 | 6.38x10 <sup>-7</sup> | -0.46 | 0.030 | 1.87x10 |
| rs1353649 | 11 | 20,253,599 | 0.99 | A/G | 0.42 | ` , | -0.03 | 0.762 | 0.19 | 0.106 | 0.215 |
| rs4980524 | 11 | 63,959,259 | 0.99 | C/A | 0.32 | STIP1 | 0.15 | 0.189 | -0.21 | 0.109 | 0.218 |
| rs6591838 | 11 | 63,959,356 | 0.99 | G/A | 0.21 | STIP1 | 0.13 | 0.336 | -0.27 | 0.117 | 0.271 |
| rs2236647 | 11 | 63,964,,605 | 0.99 | C/T | 0.29 | STIP1 | -0.02 | 0.856 | 0.03 | 0.837 | 0.975 |
| rs1144764 | 11 | 77,870,486 | 0.94 | T/C | 0.39 | KCTD21-<br>AS1 (ALG8) | 0.13 | 0.218 | -0.03 | 0.839 | 0.415 |
| rs12891009 | 14 | 74,083,846 | 0.93 | T/C | 0.27 | ACOT6/HEA<br>TR4<br>(ACOT4) | 0.31 | 0.012 | -0.36 | 0.029 | 0.026 |
| rs2230155 | 15 | 59,510,189 | 0.90 | A/G | 0.38 | MYO1É | 0.29 | 0.014 | -0.06 | 0.750 | 0.028 |
| rs12438740 | 15 | 59,515,767 | 1.00 | A/G | 0.38 | MYO1E | 0.30 | 0.012 | -0.07 | 0.699 | 0.024 |
| rs242941 | 17 | 43,892,520 | 1.00 | C/A | 0.42 | CRHR1 | -0.02 | 0.829 | 0.15 | 0.183 | 0.367 |
| rs242939 | 17 | 43,895,579 | 1.00 | C/T | 0.31 | CRHR1 | 0.04 | 0.734 | 0.13 | 0.368 | 0.433 |
| rs1876828 | 17 | 43,911,525 | 0.99 | T/C | 0.06 | CRHR1 | -0.69 | 0.007 | 0.45 | 0.026 | 0.010 |
| rs2240017 | 17 | 45,810,919 | 0.38 | G/C | 0.01 | TBX21 | -0.60 | 0.334 | 3.55 | 2.52x10 <sup>-6</sup> | 0.010 |
| rs1380657 | 17 | 48,598,785 | 1.00 | G/A | 0.13 | MYCBPAP<br>(SPATA20) | -0.16 | 0.348 | -0.13 | 0.504 | 0.262 |
| rs6504666 | 17 | 48,601,328 | 1.00 | G/A | 0.16 | MYCBPAP<br>(SPATA20) | 0.08 | 0.572 | -0.06 | 0.663 | 0.840 |
| rs9303988 | 18 | 6,667,583 | 0.67 | T/C | 0.39 | , | 0.01 | 0.948 | -0.10 | 0.438 | 0.672 |
| rs279728 | 20 | 45,080,421 | 1.00 | T/C | 0.21 | | 0.48 | 3.36x10 <sup>-4</sup> | 0.23 | 0.191 | 1.43x10 |
| rs2037925 | 21 | 40,699,931 | 0.95 | C/T | 0.37 | (BRWD1) | -0.34 | 0.003 | -0.07 | 0.538 | 0.001 |
| rs2836987 | 21 | 40,706,594 | 0.94 | C/T | 0.34 | (BRWD1) | -0.19 | 0.103 | -0.08 | 0.457 | 0.047 |
| rs138335 | 22 | 41,227,086 | 0.83 | C/G | 0.08 | ST13 | 0.19 | 0.298 | -0.22 | 0.470 | 0.575 |

rs138337 22 41,231,053 0.94 G/A 0.41 ST13 0.11 0.305 0.00 0.985 0.471

SAPPHIRE denotes Study of Asthma Phenotypes and Pharmacogenomic Interactions by Race-ethnicity; SNP, single nucleotide polymorphism; Chr, chromosome; MAF, minor allele frequency; and ICS, inhaled corticosteroid.

\*SNPs were selected from variants previously reported to be associated with ICS response. Cox proportional hazards models were used to assess associations with time-to-severe asthma exacerbation (i.e., burst oral corticosteroid use, asthma-related emergency department visits, and hospitalizations for asthma).

†The imputation quality score is the MACH-based imputation r<sup>2</sup> value, which ranges from zero to one. Values closer to one indicate higher imputation quality.

‡The "effect" allele is shown first, and the referent allele follows. The allele frequency of the "effect" allele is provided, and in the current table, this estimate is based on the observed frequency in the validation set.

§The parameter estimates represent the risk (i.e., hazard) of having a severe asthma exacerbation following the initial (baseline) assessment at study entry. A *negative* parameter estimate indicates that the variable was associated with a lower risk of experiencing a severe asthma exacerbation. The parameter estimate for the SNP can be interpreted as the effect on exacerbation risk for each additional "effect" allele (i.e., none [=0], one [=1], or two alleles [=2]). The parameter estimate for the interaction term can be interpreted as the combined effect of increasing ICS use (i.e., average number of ICS doses taken per day – see Methods Section and Supplemental Methods Section for more details on how longitudinal ICS exposure measures were created) and the number of "effect" alleles on the risk of a severe asthma exacerbation.

The P-values for the SNP and SNP x ICS interaction variables are shown for the model simultaneously including these variables, as well as adjusting for patient age, sex, BMI, smoking status, ACT score at baseline (i.e., time of study enrollment), baseline asthma severity score, LABA use (an indicator variable denoting use of an ICS-LABA combination inhaler), time-updated measures of SABA MDI and nebulizer use, the first 3 principal components, and the time-updated ICS exposure measure.

¶The likelihood ratio test assessed the significance of the difference in model fit between the full model (i.e., all of the aforementioned variables included) and the reduced model (i.e., the full model minus both the SNP and SNP x ICS interaction terms). In other words, a *joint test* was used to simultaneously assess the combined significance of the SNP and SNP x ICS interaction terms.

Table E3. Relationship between rs3827907 genotype and inhaled corticosteroid use on change in asthma control stratified by pre-treatment eosinophilia African American individuals in the SAPPHIRE cohort\*

| Sample | Sample size | rs3827907 C-all | ele status | ICS us | e | SNP*ICS interaction | |
|---|---|---|---|---|---|---|---|
| | | Parameter<br>estimate† | P-value | Parameter estimate† | P-value | Parameter estimate† | P-value |
| All | 243 | -2.569 | 5.38x10 <sup>-4</sup> | 0.097 | 0.851 | 4.405 | 1.52x10 <sup>-5</sup> |
| High EDN‡ | 121 | -3.838 | $9.87x10^{-5}$ | -0.014 | 0.984 | 5.485 | 1.35x10 <sup>-4</sup> |
| Low EDN‡ | 122 | -1.154 | 0.314 | 0.365 | 0.658 | 3.319 | 0.029 |
| High Eosinophils§ | 56 | -2.720 | 0.238 | -0.777 | 0.567 | 7.050 | 0.041 |
| Low Eosinophils§ | 57 | -2.365 | 0.154 | -0.753 | 0.533 | 3.722 | 0.075 |
| C-allele carrier | 61 | | | 4.304 | 4.61x10 <sup>-5</sup> | | |
| High EDN‡ | 28 | | | 5.986 | 0.002 | | |
| Low EDN‡ | 33 | | | 4.247 | 0.003 | | |
| High Eosinophils§ | | | | 10.234 | 0.516 | | |
| Low Eosinophils§ | | | | 2.765 | 0.116 | | |
| TT homozygotes | 182 | | | 0.14 | 0.782 | | |
| High EDN‡ | 93 | | | 0.131 | 0.830 | | |
| Low EDN‡ | 89 | | | 0.327 | 0.713 | | |
| High Eosinophils§ | 45 | | | -0.627 | 0.621 | | |
| Low Eosinophils§ | 39 | | | -1.079 | 0.415 | | |

SAPPHIRE denotes Study of Asthma Phenotypes and Pharmacogenomic Interactions by Race-ethnicity; ICS, inhaled corticosteroid; SNP, single nucleotide polymorphism; and EDN, eosinophil-derived neurotoxin.

†Parameter estimates represent the effect of a one-unit increase in the variable listed. The rs3827907 genotype was collapsed into C-allele carriers (=1) and TT homozyogotes (=0). Inhaled corticosteroid use was dichotomously categorized into those whose adherence was  $\leq$ 75% (low use) and  $\geq$ 75% (high use) over course of the 6-week treatment regimen. The interaction term represents the combined effect of rs3827907 C-allele carrier status and level of ICS use. The models used to create the parameter estimates simultaneously

<sup>\*</sup>The analysis was restricted to SAPPHIRE participants from the discovery set with available data and who underwent 6 weeks of observed ICS treatment. Change is asthma control was taken as the change in Asthma Control Test composite score from before to after ICS treatment.

included all of the variables shown, as well as variables to adjust for patient age, sex, BMI, smoking status, ACT score at baseline, and first 3 principal components. Positive parameter estimates suggest that the variable was associated with an improvement in asthma control over the 6-week ICS treatment trial.

‡The study population was stratified based on the median EDN serum level for the entire group with these data (n=243) prior to initiating ICS treatment. A baseline EDN value  $\leq$ 2.34 ng/mL was considered low and a value >2.34 ng/mL was considered high. §The study population was also stratified based on the median blood eosinophil for the entire group with these data (n=133) prior to initiating ICS treatment. A baseline blood eosinophil count  $\leq$ 222 cells/ $\mu$ L was considered low and a count >222 cells/ $\mu$ L was considered high.

(SAPPHIRE) - NCT01142947 Last updated: 02/19/2019

Table E4. Relationship between both rs3827907 and rs12891519 genotype and *RNASE2* gene expression in peripheral blood among African American participants with and without asthma from the SAPPHIRE cohort.

| Groups | rs3827907 | variant | rs12891518 variant | |
|---|---|---|---|---|
| | Parameter estimate* | P-value | Parameter estimate* | P-value |
| All participants (n=597) | -0.237 | 0.004 | -0.235 | 0.008 |
| Asthma cases (n=408) | -0.243 | 0.018 | -0.220 | 0.047 |
| Controls (n=189) | -0.224 | 0.103 | -0.267 | 0.069 |

SAPPHIRE denotes the Study of Asthma Phenotypes and Pharmacogenomic Interactions by Race-ethnicity.

\*Linear regression was used to examine the relationship between both rs3827907 genotype (coded as TT=0, CT=1, CC=2) and rs12891518 genotype (code AA=0, AT=1, and TT=2) and gene expression (dependent variable). The model adjusted for patient age, sex, BMI, the absolute cell counts for each of the 5 white blood cell types measured (i.e., neutrophils, monocytes, lymphocytes, eosinophils, and basophils from complete blood counts obtained at the time that the RNA was collected), sequence batch, and the first 30 probabilistic estimation of expression residuals (PEERs). The parameter estimates are the adjusted genotype main effect estimates for rs3827907 and rs12891518. A negative parameter estimate suggests that the minor allele (i.e., the C-allele for rs3827907 and the T-allele for rs12891518) was associated with decreased *RNASE2* gene expression.